CLINICAL TRIAL: NCT03748576
Title: Clinical Research on Mobile Medical Used for the Management of Pregnant Women: a Randomized Control Trail
Brief Title: A Prospective Randomized Controlled Trial of Mobile Medical Used for Management of Pregnant Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: JS-1012
Record Dates: First submitted 2018-10-31; First posted 2018-11-21 (Actual); Last update posted 2020-07-24 (Actual); Status verified 2018-10

CONDITIONS: Maternal Behavior; Mobile Health; Pregnancy Outcome; GDM; Blood Glucose; Diet Habit; Compliance, Patient
MeSH Terms: conditions — Feeding Behavior; Patient Compliance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mobile technologies group (Experimental): m-health group (Intervention Group) participants were managed continuously through WeChat group chat during prenatal clinic interval.
  Interventions: Behavioral: telemedicine: management through WeChat group chat
- control group (No Intervention): Standard Clinic Prenatal Care (Control Group): regular routine prenatal care following Chinese standard.

INTERVENTIONS:
Behavioral: telemedicine: management through WeChat group chat — Patients in intervention group received additional WeChat group management when conducted standard clinic prenatal care
  Arms: Mobile technologies group

SUMMARY:
A multicenter, randomized controlled trial was conducted to investigate whether health education and life style management through WeChat group chat was: 1. more effective in improving pregnancy outcomes in normal pregnant women. 2. more effective in controlling blood glucose (BG) than standard clinic prenatal care in women with GDM.

DETAILED DESCRIPTION:
1. Mobile technology and equipment based on Internet and communications technology have revolutionized the content and manner of social interaction and services. Mobile medical care has just started, the relevant platform and service is still immature, not standardized, poor satisfaction, low efficiency, its value and effectiveness of health management lack of clear theoretical support and data description. In this study, based on the multi-center prospective randomized controlled study, we constructed a large-scale maternal health service platform and a systematic standardized maternal health management model to carry out personalized maternal health management and mobile health services. Mobile medical effects validation, and further improve the mobile medical platform.

   This study will verify the value of mobile health care for maternal health management, to establish a standardized standard mobile medical model, to further improve the level of domestic maternal health management and improve the quality of maternal and child health management.
2. Most gestational diabetes mellitus (GDM) can be well controlled by health education and life style management, expecting a better pregnancy outcome. But standard clinic prenatal care which consist of clinic visit every two weeks may not give full play to the effects of GDM management. Telemedicine shows its potential to fill this gap. A multicenter, randomized controlled trial was designed to investigate whether health education and life style management through WeChat group chat was more effective in controlling blood glucose (BG) than standard clinic prenatal care in women with GDM. Women with GDM diagnosed by oral glucose tolerance test between 23-30+6 gestational weeks were randomized to a WeChat group chat-based blood glucose management group or routine clinic prenatal care. In PUMCH, investigators also equip CGM for m-health group allowing a more detailed BG information. The primary outcome was change of glycemic qualification rate during follow up period in both groups. The second outcome was pregnancy outcomes. Also, a case control study is designed to compare the glucose control status between rice-richen meal and wheaten-richen meal, and all other macronutrients and micronutrients are all calculated and same between two groups, which may provide more clues for type of carbohydrate recommendation for Chinese women with GDM.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 45 years.
* With singleton pregnancy
* Diagnosed or not diagnosed as GDM by 75g oral glucose tolerance test (OGTT) and insulin treatment is not required assessed by multi-disciplinary consultation.
* Be able to use smart phone for chatting, read and write basic Chinese.
* Volunteer for research.

Exclusion criteria:

* Pregnancies with diagnosed chronic disease
* Pregnancies with other pregnancy complications except GDM
* Pregnancies had recent trauma and treatment of glucocorticoids

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 640 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-05-31 (Actual)

PRIMARY OUTCOMES:
weight gain during pregnancy | up to 40 gestatinal weeks
  Participants record their body weight twice a month. Weight gain from third-trimester and the whole pregnancy period are calculated.
Glycemic qualification rate in women with GDM | From enrollment to 42 days postpartum
  Glycemic qualification rate was calculated by the number of BG within the control range /30*100%. BG control range were fasting BG (fasting and before-sleep BG)#95 mg/dL (5.3 mmol/L) and two-hour postprandial BG (post-breakfast, post-lunch, post-dinner BG)#120 mg/dL (6.7 mmol/L)

SECONDARY OUTCOMES:
The incidence rate of specific pregnant outcomes in both normal pregnant women and women with GDM | at delivery
  pregnancy outcomes include delivery mode, premature rupture of the membranes, preterm birth, SGA, LGA and postpartum hemorrhage

CONTACTS AND LOCATIONS:
Overall Officials: liangkun ma, Study Director — Peking union medical college hosiptal
Locations (1):
- Department of ob gyn, Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tian Y, Zhang S, Huang F, Ma L. Comparing the Efficacies of Telemedicine and Standard Prenatal Care on Blood Glucose Control in Women With Gestational Diabetes Mellitus: Randomized Controlled Trial. JMIR Mhealth Uhealth. 2021 May 25;9(5):e22881. doi: 10.2196/22881. PMID 33783365
- [Derived] Huang F, Zhang S, Tian Y, Li L, Li Y, Chen X, Sun X, Fan Y, Ma W, Liu C, Gao L, Xue X, Ma L. Effect of mobile health based peripartum management of gestational diabetes mellitus on postpartum diabetes: A randomized controlled trial. Diabetes Res Clin Pract. 2021 May;175:108775. doi: 10.1016/j.diabres.2021.108775. Epub 2021 Mar 23. PMID 33771645